CLINICAL TRIAL: NCT03747575
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Multicenter Study to Assess the Efficacy and Safety of MSTT1041A in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Assess the Efficacy and Safety of MSTT1041A in Participants With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS40965; 2018-003429-27 (EudraCT Number)
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — astegolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants will receive MSTT1041A
  Interventions: Drug: MSTT1041A
- Placebo (Placebo Comparator): Participants will receive placebo matched to MSTT1041A
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSTT1041A — Participants will receive subcutaneous (SC) MSTT1041A
  Other Names: astegolimab
  Arms: Treatment
Drug: Placebo — Participants will receive SC placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of MSTT1041A (astegolimab) in participants with moderate to severe atopic dermatitis (AD). The study consists of a screening period, a 16-week treatment period, and an 8-week follow-up period.

ELIGIBILITY:
Inclusion criteria

* Ability to comply with the study protocol
* Chronic AD that has been present for at least 3 years before the screening visit
* Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with topical medications (medications or treatments applied directly to part of the body) or for whom topical treatments are otherwise medically inadvisable

Exclusion criteria

* Prior treatment with MSTT1041A
* Treatment with any investigational therapy (with the exception of biologics) within 8 weeks or within 5 half-lives whichever is longer, before screening
* Treatment with any cell-depleting agents within 6 months before screening, or until lymphocyte count returns to normal, whichever is longer
* Treatment with other biologics within 3 months or 5 half-lives before screening, whichever is longer
* Comorbid conditions that may interfere with evaluation of investigational medicinal product
* History or evidence of substance abuse that would pose a risk to participant safety, interfere with the conduct of the study, have an impact on the study results, or affect the participant's ability to participate in the study
* History of anaphylaxis, hypersensitivity to a biologic agent, or known hypersensitivity to any component of the MSTT1041A or placebo injection
* Planned surgical intervention during the course of the study
* Pregnant or breastfeeding, or intending to become pregnant during the study
* Participant who is a member of the investigational team or his/her immediate family

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (21):
- United States (15):
  - Alabama Allergy & Asthma, Birmingham, Alabama
  - California Allergy and Asthma Medical Group - CRN, Los Angeles, California
  - Jonathan Corren MD, Inc., Los Angeles, California
  - Asthma & Allergy; Associates, P.C., Colorado Springs, Colorado
  - South Coast Research Center, Inc., Miami, Florida
  - Harmony Clinical Research, Inc, North Miami Beach, Florida
  - GCP Global Clinical Professionals, St. Petersburg, Florida
  - Forward Clinical Trials, Tampa, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Midwest Sinus Allergy and Asthma - CRN, Normal, Illinois
  - Dermatology Specialists Research, LLC, Louisville, Kentucky
  - Clinical Research Consortium Nevada, Las Vegas, Nevada
  - Skin Laser and Surgery Specialists of New York and New Jersey LLC - Interspond - PPDS, Hackensack, New Jersey
  - Vital Prospects Clinical Research Institute PC - CRN, Tulsa, Oklahoma
  - Center for Clinical Studies, Houston, Texas
- Universitatsklinikum Munster, Münster, Germany
- Poland (5):
  - Centrum Medyczne ALL-MED, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Kliniczny Szpital Wojewodzki Nr 1 im. Fryderyka Chopina; Klinika Dermatologii, Rzeszów
  - Laser Clinic, Szczecin
  - Wro Medica, Wroc?aw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com).
  Further details on Roche's criteria for eligible studies are available here: https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here: (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received a loading dose of SC placebo matched to MSTT1041A followed by SC placebo Q4W.
- Treatment: Participants received a loading dose of 245 mg of subcutaneous (SC) MSTT1041A, followed by 490 mg of SC MSTT1041A every 4 weeks (Q4W).
Period: Overall Study
Arm/Group | Placebo | Treatment
Started | 32 | 33
Completed | 23 | 26
Not Completed | 9 | 7
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 31 | 61
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (14.4) | 39.7 (15.2) | 39.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 20 | 25 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Total Eczema Area and Severity Index (EASI) Score
Description: The Eczema Area and Severity Index (EASI) is a standardized instrument to evaluate the extent and severity of atopic dermatitis. An area score comprised of the percentage of skin affected by eczema for each of 4 body regions (head/neck, trunk, upper extremities, and lower extremities) is calculated with 0 = none, 1 = 1-9%, 2 = 10-29%, 3 = 30-49%, 4 = 50-69%, 5 = 70-89%, and 6 = 90-100%. Severity is scored for each of the 4 body regions by the summation of the intensity scores for 4 signs (redness, thickness, scratching, and lichenification), with 0 = none/absent, 1 = mild, 2 = moderate, and 3 = severe. The minimum final EASI score is 0 and the maximum score is 72.
Time Frame: Baseline, Week 16
Population: ITT population - all participants randomized on Day 1, grouped by the treatment assigned at randomization.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 32
Percentage | -51.47 (8.639) | -58.24 (9.092)

2. Secondary Outcome: Proportion of Participants Who Achieve Investigator's Global Assessment (IGA) Response of 0 or 1
Time Frame: Baseline, Week 16
Population: ITT population - all participants randomized on Day 1, grouped by the treatment assigned at randomization.
Measure: Number; unit: Percentage
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 32
Percentage | 15.2 | 6.3

3. Secondary Outcome: Proportion of Participants Who Achieve >/=75% Reduction From Baseline in Eczema Area and Severity Index (EASI-75) Score
Time Frame: Baseline, Week 16
Population: ITT population - all participants randomized on Day 1, grouped by the treatment assigned at randomization.
Measure: Number; unit: Percentage
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 32
Percentage | 27.3 | 18.8

4. Secondary Outcome: Percent Change in Pruritus as Assessed by a Numeric Rating Scale (NRS)
Description: The Peak Pruritis Numerical Rating Scale (NRS) is a single-item patient-reported outcome (PRO) of itch severity rated on a scale of 0-10, with 0 = no itch and 10 = worst itch imaginable for the prior 24-hour period.
Time Frame: Baseline, Week 16
Population: ITT population - all participants randomized on Day 1, grouped by the treatment assigned at randomization.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 32
Percentage | -31.22 (7.376) | -39.43 (7.839)

5. Secondary Outcome: Percent Change in Body Surface Area (BSA) With Atopic Dermatitis (AD) Involvement
Time Frame: Baseline, Week 16
Population: ITT population - all participants randomized on Day 1, grouped by the treatment assigned at randomization.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 32
Percentage | -42.23 (8.637) | -38.87 (9.134)

6. Secondary Outcome: Percent Change in Disease Severity as Assessed by SCORing Atopic Dermatitis (SCORAD)
Description: SCORAD is a tool used to assess the extent and severity of eczema based on three aspects of disease severity: extent, intensity, and a subjective (PRO) symptoms. A total score (0-103) is calculated, with higher scores indicating a higher extent and severity of symptoms.
Time Frame: Baseline, Week 16
Population: ITT population - all participants randomized on Day 1, grouped by the treatment assigned at randomization.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 32
Percentage | -35.45 (6.837) | -39.50 (7.202)

7. Secondary Outcome: Percentage of Participants With Adverse Events (AE)
Time Frame: Up to Week 24
Population: Safety population - all randomized participants who received at least one dose of study drug. Participants are grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 34 | 31
Participants | 14 | 18

8. Secondary Outcome: Serum Concentrations of MSTT1041A
Time Frame: At pre-defined intervals from baseline up to Week 24
Population: PK population: The PK population included participants from the safety population with at least one available post-study treatment PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Treatment
Number analyzed (Participants) | 33
ug/mL
  Day 1 Visit 2/prior to infusion: number analyzed (Participants) | 32
  Day 1 Visit 2/prior to infusion | NA (NA) — Summary statistics are not reportable for sampling time points in which more than one-third of the samples were less than reportable (LTR; the value of LTR was set to zero).
  Week 1 Visit 3/prior to infusion | 42.6 (34.4)
  Week 4 Visit 5/prior to infusion | 37.6 (52.5)
  Week 8 Visit 7/prior to infusion: number analyzed (Participants) | 28
  Week 8 Visit 7/prior to infusion | 36.6 (54.5)
  Week 12 Visit 9/prior to infusion: number analyzed (Participants) | 26
  Week 12 Visit 9/prior to infusion | 40.1 (60.5)
  Week 16 Visit 11: number analyzed (Participants) | 26
  Week 16 Visit 11 | 38.2 (76.0)
  Subject disposition - period completion/early discontinuation: number analyzed (Participants) | 26
  Subject disposition - period completion/early discontinuation | 7.83 (151.2)

9. Secondary Outcome: Incidence of Treatment-Emergent Anti-Drug Antibodies (ADAs)
Time Frame: Up to Week 24
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 34 | 31
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: The safety population contained all randomized participants who received at least one dose of study drug. Participants are grouped according to actual treatment received.
Arm/Group | Placebo | Treatment
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/34
Other Adverse Events (participants affected / at risk) | 8/31 | 3/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Treatment (N=34)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Treatment (N=34)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (5) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT03747575/Prot_SAP_000.pdf